CLINICAL TRIAL: NCT02869451
Title: Mobile Contingency Management for Concurrent Abstinence From Cannabis and Cigarette Smoking: A Pilot Study
Brief Title: Mobile Contingency Management for Marijuana and Tobacco Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00072366
Record Dates: First submitted 2016-08-08; First posted 2016-08-17 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Cigarette Smoking; Marijuana Abuse
MeSH Terms: conditions — Cigarette Smoking; Marijuana Abuse | interventions — Bupropion; Tobacco Use Cessation Devices; Nicotine Chewing Gum; Counseling; nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Cognitive-behavioral counseling for marijuana and smoking cessation, mobile contingency management for marijuana and smoking cessation, transdermal nicotine patch (7-21 mg over six weeks), nicotine polacrilex or nicotine lozenge (4 mg administered as needed over six weeks), bupropion (150 mg once per day for 7 days, then 150 mg twice per day for about six months.
  Interventions: Drug: bupropion; Drug: transdermal nicotine patch; Drug: Nicotine polacrilex; Drug: nicotine lozenge; Behavioral: counseling for marijuana and smoking cessation; Behavioral: mobile contingency management

INTERVENTIONS:
Drug: bupropion — Prescribed one week prior to quit and continued until the 6 month follow-up visit.
  Other Names: Zyban
Drug: transdermal nicotine patch — Initiated at smoking quit date; 7 mg to 21 mg patch depending on amount smoked by participant
Drug: Nicotine polacrilex — Initiated at smoking quit date.
  Other Names: nicotine gum; nicorette
Drug: nicotine lozenge — Initiated at smoking quit date.
Behavioral: counseling for marijuana and smoking cessation — 5 sessions of cognitive-behavioral counseling designed to facilitate marijuana and smoking cessation and promote relapse prevention
Behavioral: mobile contingency management — treatment that provides money rewards for abstinence from smoking and marijuana

SUMMARY:
The purpose of this pilot project is to pilot-test a combined cannabis and smoking cessation treatment. The intervention combines mobile technology with behavioral strategies, counseling, and medications.

DETAILED DESCRIPTION:
Cannabis is the most widely used illicit drug in the United States with 19.8 million current users. Population based data indicate that almost all cannabis users (90%) have a lifetime history of tobacco smoking and the majority (74%) currently smoke tobacco. While cannabis use alone is associated with significant adverse health effects, tobacco smoking is the number one preventable cause of illness and death in the U.S. This is true even among those using illicit drugs where the tobacco -related mortality rate is twice that of the general population. Among cannabis users, smoking tobacco is associated with increased frequency of marijuana use, increased morbidity, and poorer cannabis cessation outcomes. There is strong evidence for the short -term efficacy for cannabis use disorder (CUD) and smoking of contingency management (CM). It is an intensive behavioral therapy that provides incentives (vouchers, money) to individuals misusing substances contingent upon objective evidence from drug use. Implementation of CM has been limited because of the need to verify abstinence multiple times daily using clinic based monitoring and effects are short lived. The investigators recently developed a smart -phone application which allows a patient to video themselves several times daily while using a small CO monitor and to transmit the data to a secure server which has made the use of CM for outpatient smoking cessation portable and feasible. The mobile CM (mCM) approach paired with cognitive-behavioral counseling and pharmacological smoking cessation aids has been effective in reducing smoking in the short and long-term. The purpose of this pilot project is to pilot-test a combined cannabis and smoking mCM intervention. The pilot will allow the investigators to examine feasibility of the treatment and of planned recruitment strategies. These project aims will provide the first step toward implementation of an innovative approach that builds upon the power of mHealth technology to reduce the prevalence of both CUD and cigarette smoking.

ELIGIBILITY:
Inclusion Criteria:

* report 40 or more days of cannabis use in the past 90 day;
* have smoked at least seven cigarettes in the past seven days;
* have been smoking for at least the past year;
* can speak and write fluent conversational English;
* are between 18 and 70 years of age; and
* are willing to make an attempt to quit both cannabis and tobacco smoking.

Exclusion Criteria:

* expected to have unstable medication regimen during the study;
* currently receiving non-study behavioral treatment for cannabis use disorder or smoking;
* myocardial infarction in past six months;
* contraindication to NRT with no medical clearance;
* use of other forms of nicotine such as cigars, pipes, or chewing tobacco with unwillingness to stop use of these forms;
* current pregnancy;
* primary psychotic disorder or current manic episode;
* substance use disorder (other than cannabis or nicotine) within the preceding three months; or
* current imprisonment or psychiatric hospitalization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean C Beckham, Ph.D., Principal Investigator — Study Principal Investigator
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment occurred between August 2016 to May 2017. Participants were recruited from community settings and Craigslist.
Pre-assignment Details: Seven participants signed consent. Two of these participants were withdrawn by the principal investigator after signing consent because they did not meet study eligibility criteria.
Period: Overall Study
Arm/Group | Treatment
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Self-report Prolonged Abstinence From Smoking
Description: Participants self-report smoking behavior since smoking quit date. Prolonged abstinence is defined as sustained abstinence since two weeks post-initial smoking quit date.
Time Frame: 6 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 0

2. Primary Outcome: Number of Participants Who Report Smoking Abstinence and Abstinence is Bioverified by Salivary Cotinine
Description: Self-reported abstinence (primary outcome) will be verified by cotinine assay. Saliva samples will be collected from participants who self-report prolonged abstinence.
Time Frame: 6 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 0

3. Primary Outcome: Number of Participants Who Self-report Prolonged Abstinence From Marijuana Use
Description: Participants self-report marijuana use since marijuana quit date. Prolonged abstinence is defined as sustained abstinence since two weeks post-initial quit date.
Time Frame: 6 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 0

4. Primary Outcome: Number of Participants Who Report Marijuana Abstinence and Abstinence is Bioverified by Oral Fluid
Description: Self-reported abstinence (primary outcome) will be verified by oral fluid (OF) cannabis assessment. Oral fluid samples will be collected from participants who self-report prolonged abstinence.
Time Frame: 6 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 0

5. Secondary Outcome: Number of Participants Who Self-report 7 Day Point Prevalence Abstinence From Smoking
Description: 7-day point prevalence abstinence is defined as no smoking in the prior 7 days.
Time Frame: 6 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 1

6. Secondary Outcome: Number of Participants Who Self-report 7 Day Point Prevalence Abstinence From Marijuana
Description: 7-day point prevalence abstinence is defined as no marijuana use in the prior 7 days.
Time Frame: 6 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 2

7. Secondary Outcome: Number of Participants Who Report 30 Day Point Prevalence Abstinence From Marijuana
Description: 30-day point prevalence abstinence is defined as no marijuana use in the prior 30 days.
Time Frame: 6 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 1

8. Secondary Outcome: Number of Participants Who Report 30 Day Point Prevalence Abstinence From Smoking
Description: 30-day point prevalence abstinence is defined as no smoking in the prior 30 days.
Time Frame: 6 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 1

9. Secondary Outcome: Number of Participants Who Report 7 Day Point Prevalence Abstinence From Smoking
Description: 7-day point prevalence abstinence is defined as no smoking in the prior 7 days.
Time Frame: 3 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 0

10. Secondary Outcome: Number of Participants Who Report 7 Day Point Prevalence Abstinence From Marijuana
Description: 7-day point prevalence abstinence is defined as no marijuana use in the prior 7 days.
Time Frame: 3 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 3

11. Secondary Outcome: Number of Participants Who Report Smoking Abstinence and Abstinence is Bioverified by Salivary Cotinine
Description: as for outcome 2
Time Frame: 3 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 0

12. Secondary Outcome: Number of Participants Who Report Marijuana Abstinence and Abstinence is Bioverified by Salivary Cotinine
Description: as for outcome 4
Time Frame: 3 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 3

13. Secondary Outcome: Change From Baseline in Number of Days Per Week of Cannabis Use
Description: Participants will self-report amount of marijuana used in past week; this will be compared to self-reported amount smoked per week prior to quit date.
Time Frame: baseline, 6 month follow up
Measure: Mean (Standard Deviation); unit: days per week of marijuana use
Arm/Group | Treatment
Number analyzed (Participants) | 5
days per week of marijuana use | -3.4 (1.34)

14. Secondary Outcome: Proportional Change in Days of Cannabis Use From Pre-quit to 6 Month Follow-up (Entire Group)
Description: Participants will self-report number of days marijuana used in the past 30 days and this will be compared for the entire group to self-reported number of days of use in 30 days prior to quit. The proportion will be calculated by totaling baseline days used and pretreatment days used, and then dividing baseline days used by pretreatment days used.
Time Frame: 30 days prior to quit date, 6 month follow up
Measure: Number; unit: percentage of pre-quit use
Arm/Group | Treatment
Number analyzed (Participants) | 5
percentage of pre-quit use | 28

15. Secondary Outcome: Change in Number of Cigarettes Smoked Per Week Compared to Pre-quit
Description: Self-reported number of cigarettes smoked each day in past 7 days; this will be compared to self-reported amount smoked in week prior to quit date
Time Frame: 7 days prior to quit date, 6 month follow up
Measure: Mean (Standard Deviation); unit: number of cigarettes per wk
Arm/Group | Treatment
Number analyzed (Participants) | 5
number of cigarettes per wk | -37.8 (39.16)

16. Secondary Outcome: Proportional Change in Days Smoked From Pre-quit to 6-month Follow up (for Entire Group)
Description: Participants will self-report number of days smoked in the past 30 days and this will be compared (for the entire group) to self-reported number of days smoked in 30 days prior to quit. The proportion will be calculated by totaling baseline days used and pretreatment days used, and then dividing baseline days used by pretreatment days used.
Time Frame: 30 days prior to quit date, 6 month follow up
Measure: Number; unit: percentage of pre-quit use
Arm/Group | Treatment
Number analyzed (Participants) | 5
percentage of pre-quit use | 80

17. Secondary Outcome: Percentage of Missing Mobile Contingency Management Video Recordings
Description: Participants upload video recordings of abstinence verification as part of contingency management treatment. Percentage of missed videos (compared to expected videos) will be assessed as a measure of feasibility of the contingency management intervention
Time Frame: 3 month follow up
Measure: Number; unit: percent missed video recordings
Arm/Group | Treatment
Number analyzed (Participants) | 5
percent missed video recordings | 33.9

18. Secondary Outcome: Number of Missed Behavioral Counseling Sessions
Description: Participants attend telephone counseling sessions. Number of missed sessions for the total group will be assessed as a measure of acceptability of the behavioral counseling
Time Frame: 3 month follow up
Measure: Number; unit: missed counseling sessions
Arm/Group | Treatment
Number analyzed (Participants) | 5
missed counseling sessions | 0

19. Secondary Outcome: Number of Voluntary Withdrawals From the Project
Description: The number of participants who withdraw from the study will be evaluated as a measure of treatment feasibility and acceptability
Time Frame: Evaluated at 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for approximately seven months, from informed consent signature to 6-month follow-up (which occurred 6 months after substance cessation date).
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=5)
Nausea with bupropion use (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT02869451/Prot_SAP_ICF_000.pdf